CLINICAL TRIAL: NCT02670278
Title: Evolutionary and Sociocultural Aspects of Human Milk Composition
Acronym: INSPIRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Other Study IDs: 24300409
Record Dates: First submitted 2016-01-20; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — milk, feces, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (11):
- US-Washington, Idaho: healthy breastfeeding women and their infants
- US-California: healthy breastfeeding women and their infants
- Sweden: healthy breastfeeding women and their infants
- Spain: healthy breastfeeding women and their infants
- Peru: healthy breastfeeding women and their infants
- Kenya: healthy breastfeeding women and their infants
- Ethiopia-rural: healthy breastfeeding women and their infants
- Ethiopia-urban: healthy breastfeeding women and their infants
- The Gambia-rural: healthy breastfeeding women and their infants
- The Gambia-urban: healthy breastfeeding women and their infants
- Ghana: healthy breastfeeding women and their infants

SUMMARY:
It is well-known that breastfeeding protects infants from illness, especially in the poorest regions of the world. The full nature of this protective effect, however, is less well understood. A major barrier to understanding is the fact that almost nothing is known about the factors that influence the considerable variation in milk composition around the globe, or about the effects of this variation on infant health. This INSPIRE project represents the first comprehensive investigation of the global differences in human milk composition along with the various microbial, evolutionary, environmental, and sociocultural factors that might influence both milk composition and infant health. An international, interdisciplinary collaboration of physiologists, nutritional scientists, anthropologists, microbiologists, and mathematicians will collect biological data from breastfeeding women and their infants, in concert with extensive anthropologic and ecological data, in both developed (US, Spain, Sweden) and developing countries (Central African Republic, Gambia, Ghana, Peru, and Kenya). To test the possibility of a correlation between milk oligosaccharide composition, milk microbiota, and the gastrointestinal microbiome of infants, milk samples and infant fecal samples will be analyzed using state-of-the-art biochemical and genomic techniques. This study will allow important cross-cultural comparisons of milk composition and infant feeding practices; it also will utilize sophisticated computational methods to integrate the extensive, diverse body of combined biological and anthropological data to elucidate the relationships among sociocultural factors, evolutionary history, environmental exposures, microbial constituents and milk composition. The researchers predict that what is considered "normal" milk composition in one population may not support optimal health in another. This information is crucial to the humanitarian quest to understand how infant nutrition and overall health can be improved around the world. In addition, this project will provide extensive research training opportunities for undergraduate, graduate and postdoctoral scientists.

ELIGIBILITY:
Inclusion Criteria

* Breastfeeding or pumping at least 5 times daily (to assure adequate milk production)
* Self-reported healthy women and infants
* ≥ 18 yr of age (maternal)
* 1-3 mo postpartum

Exclusion Criteria

* Current indication of breast infection (e.g., breast pain, discomfort, lumps, mastitis with fever, red streaks, or hard red portions of the breast)
* Breast pain that the woman does not consider "normal" for lactation/breastfeeding
* Any antibiotics to mother or infant in the previous month (30 days)
* Infant has had signs/symptoms of acute illness in the previous 7 days including the following: fever, diarrhea (≥ 3 excessively "loose" stools in a day), vomiting not associated with feeding, severe cough, rapid breathing

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy breastfeeding women and their infants
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Microbial community structure of milk | 1-3 months postpartum
  Sequencing of microbial 16S gene via MiSeq; data will be analyzed as relative abundances of bacteria from phylum to genus; how milk microbial profiles are related to milk oligosaccharide and infant fecal microbiomes will be explores using multivariate ecological analyses.

SECONDARY OUTCOMES:
Sociocultural data of women, including dietary intake patterns and microbial exposures | 1-3 months postpartum
  Collected via surveys; multivariate analysis will be conducted to relate these factors to variation in primary outcomes - particularly microbial community structure of milk.
Microbial community structure of infant feces | 1-3 months of life
  Sequencing of microbial 16S gene via MiSeq; data will be analyzed as relative abundances of bacteria from phylum to genus; relationships with milk microbiome and oligosaccharide profiles will be explored using multivariate ecological analyses.
Oligosaccharide profiles of milk | 1-3 months postpartum
  Total and individual oligosaccharide concentrations will be determined; how oligosaccharide profiles are related to milk and infant microbiomes will be explores using multivariate ecological analyses.

OTHER OUTCOMES:
Maternal genomic variation related to via SNP analysis and/or genome-wide association studies | 1-3 months postpartum
  Funding not yet obtained; when garnered, we will explore relationships between maternal genomics and milk oligosaccharide profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle K McGuire, PhD, Principal Investigator — Washington State University
Locations (1):
- School of Biological Sciences, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz L, Alba C, Garcia-Carral C, Jimenez EA, Lackey KA, McGuire MK, Meehan CL, Foster J, Sellen DW, Kamau-Mbuthia EW, Kamundia EW, Mbugua S, Moore SE, Prentice AM, Gindola K D, Otoo GE, Pareja RG, Bode L, McGuire MA, Williams JE, Rodriguez JM. Comparison of Two Approaches for the Metataxonomic Analysis of the Human Milk Microbiome. Front Cell Infect Microbiol. 2021 Mar 25;11:622550. doi: 10.3389/fcimb.2021.622550. eCollection 2021. PMID 33842385
- [Derived] Ruiz L, Espinosa-Martos I, Garcia-Carral C, Manzano S, McGuire MK, Meehan CL, McGuire MA, Williams JE, Foster J, Sellen DW, Kamau-Mbuthia EW, Kamundia EW, Mbugua S, Moore SE, Kvist LJ, Otoo GE, Lackey KA, Flores K, Pareja RG, Bode L, Rodriguez JM. What's Normal? Immune Profiling of Human Milk from Healthy Women Living in Different Geographical and Socioeconomic Settings. Front Immunol. 2017 Jun 30;8:696. doi: 10.3389/fimmu.2017.00696. eCollection 2017. PMID 28713365
- [Derived] McGuire MK, Meehan CL, McGuire MA, Williams JE, Foster J, Sellen DW, Kamau-Mbuthia EW, Kamundia EW, Mbugua S, Moore SE, Prentice AM, Kvist LJ, Otoo GE, Brooker SL, Price WJ, Shafii B, Placek C, Lackey KA, Robertson B, Manzano S, Ruiz L, Rodriguez JM, Pareja RG, Bode L. What's normal? Oligosaccharide concentrations and profiles in milk produced by healthy women vary geographically. Am J Clin Nutr. 2017 May;105(5):1086-1100. doi: 10.3945/ajcn.116.139980. Epub 2017 Mar 29. PMID 28356278
- [Derived] McGuire MK, McGuire MA, Price WJ, Shafii B, Carrothers JM, Lackey KA, Goldstein DA, Jensen PK, Vicini JL. Glyphosate and aminomethylphosphonic acid are not detectable in human milk. Am J Clin Nutr. 2016 May;103(5):1285-90. doi: 10.3945/ajcn.115.126854. Epub 2016 Mar 30. PMID 27030536